CLINICAL TRIAL: NCT05438628
Title: Preoperative Frailty Assessment With Point-of-care Ultrasound in Elderly Patients Scheduled for Total Knee Arthroplasty
Brief Title: Preoperative Frailty Assessment With Ultrasound in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: 2206-089-1332
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients scheduled for total knee arthroplasty surgery
  Interventions: Diagnostic Test: Point of care ultrasound

INTERVENTIONS:
Diagnostic Test: Point of care ultrasound — Measurement of thickness of rectus abdominis, biceps brachii muscles

SUMMARY:
In this study, the investigators aim to evaluate the prediction accuracy of the thickness measured with point-of-care ultrasound of the rectus abdominis, biceps brachii muscles of frailty.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years old or older scheduled for total knee arthroplasty

Exclusion Criteria:

* Unable to communicate with the patient or the patient's guardian
* Myopathy
* History of injury of rectus abdominis, biceps brachii or quadriceps femoris muscle.
* History of total knee arthroplasty in the recent 3 months prior to surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 60 years old or older scheduled for total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Prediction accuracy of the thickness of rectus abdominis, biceps brachii muscles measured with point of care ultrasound | Preoperative evaluation

SECONDARY OUTCOMES:
Thickness of quadratus femoris muscle measured with point-of care ultrasound | Preoperative evaluation
Circumference of thigh | Preoperative evaluation
Difference between thickness of left and right rectus abdominis muscles | Preoperative evaluation
Difference between thickness of left and right biceps brachii muscles | Preoperative evaluation
Difference between thickness of left and right quadriceps femoris muscles | Preoperative evaluation
Unplanned ICU admission | First 30 days post surgery
Unplanned discharge to nursing facility | First 30 days post surgery
Incidence of postoperative delirium | First 30 days post surgery
ICU stay duration | First 30 days post surgery
Total length of stay | First 30 days post surgery
Number of falls | First 30 days post surgery
Readmission in the 30-day postoperative period | First 30 days post surgery
Mortality | First 30 days post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided